CLINICAL TRIAL: NCT02881255
Title: Avoid Transvenous Leads in Appropriate Subjects
Acronym: ATLAS S-ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATLAS S-ICD
Record Dates: First submitted 2016-08-02; First posted 2016-08-26 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Ventricular Arrhythmia
Keywords: implantable cardioverter defibrillator; subcutaneous ICD; transvenous ICD; inherited arrhythmia syndrome
MeSH Terms: interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Subcutaneous ICD (Other): Patient will receive a subcutaneous implantable cardioverter defibrillator (Boston Scientific EMBLEM)
  Interventions: Device: Implantable Cardioverter Defibrillator
- Transvenous ICD (Other): Patient will receive a single-chamber, transvenous implantable cardioverter defibrillator (from any manufacturer) which as the capability for remote monitoring.
  Interventions: Device: Implantable Cardioverter Defibrillator

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator — Patients will be randomized to receive either a subcutaneous or transvenous ICD.

SUMMARY:
The purpose of the study is to compare standard, single chamber transvenous ICD to sub-cutaneous ICD in occurrence of perioperative and long term device related complications and failed appropriate clinical shocks and arrhythmic death.

ELIGIBILITY:
Inclusion Criteria: patient must satisfy any ONE of the following two criteria:

1. Patient is ≥ 18 - 60 years old AND has a standard indication for ICD; OR
2. Patient is ≥ 18 years old AND has any one of the following present:

   * An inherited arrhythmia syndrome (i.e. Long QT, Brugada, ARVC, hypertrophic or dilated cardiomyopathy, early repolarization syndrome, idiopathic ventricular fibrillation, etc.)
   * Prior pacemaker or ICD removal for infection
   * Need for hemodialysis
   * Prior heart valve surgery (repair or replacement)
   * Chronic obstructive pulmonary disease (with FEV1 < 1.5 L)

Exclusion Criteria:

* Mechanical tricuspid valve
* Fontan repair
* Presence of an intra-cardiac shunt
* Known lack of upper extremity venous access
* Need for cardiac pacing for bradycardia indication
* PR interval of > 240 msec
* Patients with permanent pacemaker
* Clinical indication for biventricular pacing
* Patients unwilling to provide informed consent or comply with follow-up
* Pregnant at time of enrollment and implant
* Patients who currently have a ventricular assist device (i.e. LVAD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Composite of lead-related perioperative complications | 6 months post-ICD implantation
  This composite includes:
  Hemothorax or pneumothorax; Cardiac perforation, tamponade, pericardial effusion or pericarditis; Lead dislodgement or loss of pacing/sensing requiring revision; New moderate-severe or severe tricuspid insufficiency (3+ or 4+); Ipsilateral upper extremity deep venous thrombosis.
Additional safety composite | 6 months post-ICD implantation
  This composite includes:
  Device-related infection requiring surgical revision; Significant wound hematoma (requiring evacuation or interruption of oral anticoagulation); Myocardial infarction; Stroke; Death;

SECONDARY OUTCOMES:
Late device-related complications | Greater than 6 months post-ICD implantation
  The following complications will be measured by their presence or absence; they will be presented as individual complications and also as a composite of late device-related complications:
  * Lead dislodgement or fracture; or loss of adequate sensing or pacing
  * Device-related infection
  * Pericarditis or pericardial effusion
  * New severe tricuspid insufficiency
  * Ipsilateral upper extremity deep venous thrombosis
  * Need to revise dialysis access
  * Need to revise ICD or lead for any reason
  * Non-systemic embolism
  * Pulmonary embolism
  * Wound dehiscence or disjunction
  * Allergic reaction to ICD
Total device-related complications | Greater than 6 months post-ICD implantation
  This is a composite of:
  all components of the primary and secondary safety outcomes, and late device-related complications.
Occurrence of failed appropriate shock or arrhythmic death | 6 months post-ICD implantation
  Efficacy outcome
Hospital, emergency department or clinic visits for ICD therapy, device-related complications, arrhythmia or heart failure | 6 months post-ICD implantation
  Efficacy outcome. Hospital, emergency department or clinic visits for ICD therapy (shocks or anti-tachycardia pacing, both appropriate and inappropriate), device-related complications, arrhythmia or heart failure
Any inappropriate ICD therapy shock | 6 months post-ICD implantation
  Efficacy outcome
All-cause mortality | 6 months post-ICD implantation
  Efficacy outcome
Provincial healthcare payer health economics analysis | 6 months post-ICD implantation
  A formal health economics analysis will be completed as part of this study, using the perspective of a provincial healthcare payer. Procedural costs will be obtained from the Ontario schedule of benefits and the cost of device-implantation will be taken from existing, local case-costing data. The cost-effectiveness analysis will take into consideration any differences in survival, complication rates and resource utilization. Sensitivity analyses will be done, varying the price of the S-ICD, in order to generate cost-acceptability curves.
Patient Acceptance of ICD as measured by Florida Patient Acceptance Survey (FPAS) | 1 month and 6 month post-ICD implantation
  Patient acceptance of ICD will be measured using the Florida Patient Acceptance Survey (FPAS).
Patient Health Survey as measured by Short Form Health Survey (SF36) | Baseline and 6 months post-ICD implantation
  Patient health will be assessed by a generic instrument, the Short Form Health Survey (SF36). This survey provides scores for each of the eight health domains and psychometrically-based physical component summary and mental component summary scores.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Healey, MD, Principal Investigator — Population Health Research Institute; Blandine Mondesert, MD, Principal Investigator — Université de Montréal
Locations (14):
- Canada (14):
  - University of Calgary, Calgary, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario
  - IUCPQ-Universite Laval, Laval, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mondesert B, Bashir J, Philippon F, Dubuc M, Amit G, Exner D, Joza J, Birnie DH, Lane C, Tsang B, Korley V, Spears D, Ling A, Djuric A, Crystal E, Hruczkowski T, Roux JF, Carroll S, Essebag V, Krahn AD, Healey JS. Rationale and design of the randomized prospective ATLAS study: Avoid Transvenous Leads in Appropriate Subjects. Am Heart J. 2019 Jan;207:1-9. doi: 10.1016/j.ahj.2018.09.008. Epub 2018 Oct 9. PMID 30399474
- [Derived] Carroll SL, Mondesert B, Krahn AD, Bashir JG, Fisher K, Nair K, Healey JS. Device-specific quality of life: results from the ATLAS trial-avoid transvenous leads in appropriate subjects. Eur J Cardiovasc Nurs. 2024 Dec 16;23(8):877-885. doi: 10.1093/eurjcn/zvae067. PMID 38695087
- [Derived] Healey JS, Krahn AD, Bashir J, Amit G, Philippon F, McIntyre WF, Tsang B, Joza J, Exner DV, Birnie DH, Sadek M, Leong DP, Sikkel M, Korley V, Sapp JL, Roux JF, Lee SF, Wong G, Djuric A, Spears D, Carroll S, Crystal E, Hruczkowski T, Connolly SJ, Mondesert B; ATLAS Investigators. Perioperative Safety and Early Patient and Device Outcomes Among Subcutaneous Versus Transvenous Implantable Cardioverter Defibrillator Implantations : A Randomized, Multicenter Trial. Ann Intern Med. 2022 Dec;175(12):1658-1665. doi: 10.7326/M22-1566. Epub 2022 Nov 8. PMID 36343346